CLINICAL TRIAL: NCT01993030
Title: Randomized, Active-controlled, Single-blind, Parallel Two-group Trial of HQ® Matrix Medical Wound Dressing and Sidaiyi® Wound Dressing for the Treatment of Donor Site Wounds
Brief Title: Evaluation of HQ® Matrix Medical Wound Dressing for Healing of Donor Site Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Xingyue Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XY-201301
Record Dates: First submitted 2013-11-14; First posted 2013-11-25 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Donor Site Wound

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HQ® Matrix Medical Wound Dressing (Experimental): After harvesting the graft, the donor site wounds were treated with the dressing material. Dressing changes if needed. An operative removal of the HQ® Matrix Medical Wound Dressing is not required as it becomes spontaneously detached from the regenerated skin areas.
  Interventions: Device: HQ® Matrix Medical Wound Dressing
- Sidaiyi® wound dressing (Active Comparator): After harvesting the graft, the donor site wounds were treated with the dressing material. Dressing changes if needed.
  Interventions: Device: Sidaiyi® wound dressing

INTERVENTIONS:
Device: HQ® Matrix Medical Wound Dressing
  Other Names: HQ® Matrix
  Arms: HQ® Matrix Medical Wound Dressing
Device: Sidaiyi® wound dressing
  Other Names: Sidaiyi®
  Arms: Sidaiyi® wound dressing

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of HQ® Matrix Medical Wound Dressing for repair of donor site wounds. Half of participants will receive HQ® Matrix Medical Wound Dressing, while the other half will receive Sidaiyi® wound dressing.

DETAILED DESCRIPTION:
HQ® Matrix Medical Wound Dressing is a transparent, non-porous, pliable, gas-permeable, and waterproof film dressing which is comprised of silk fibroin protein of the Bombyx mori (B. mori) silkworm. It is intended to provide a moist, gas-permeable and sterile environment to facilitate the normal wound healing process. It is used in the management of non-infected skin defects and various dermal wounds.

Sidaiyi® wound dressing (Suzhou Soho Biomaterial Science and Technology Co., Ltd, Suzhou, China) is a CFDA approved (Su2012-2640182), silk fibroin-based, two-layered spongy dressing. Upon the silk fibroin spongy dressing layer is a membrane made of medical silicone. It is used in the management of partial- and full-thickness wounds, donor site wounds and burns. Currently, it is the sole silk fibroin biomaterial for wound healing that has received regulatory approval worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, aged from 18 - 60, male or female, with wet wounds or burns, ulcerative skin and soft tissue wound surfaces;
2. The wound surface area ranged from 20cm^2 to 600cm^2;
3. The patients had a clear mind and there was no misunderstanding;
4. The patients voluntarily signed the subjects' informed consent form and received timely follow-ups.

Exclusion Criteria:

1. Patients with active bleeding in wound surfaces;
2. Vasogenic diseases: patients with no blood supply or phlebothrombosis in local wound tissues;
3. Those allergic to silk materials;
4. Those with serious infection;
5. Those with coagulation disorders;
6. Those with tumors or diabetes;
7. Patients who, according to other doctors' opinion, are unsuitable to use this material for wound treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Qian, PhD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (2):
- China (2):
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan

RESULTS

PARTICIPANT FLOW:
Groups:
- HQ® Matrix Medical Wound Dressing: Dressing indicated for donor site wounds. Dressing changes every 2-3 days, more frequently if needed
  HQ® Matrix Medical Wound Dressing
- Sidaiyi® Wound Dressing: Dressing indicated for donor site wounds. Dressing changes every 2-3 days, more frequently if needed
  Sidaiyi® wound dressing
Period: Overall Study
Arm/Group | HQ® Matrix Medical Wound Dressing | Sidaiyi® Wound Dressing
Started | 36 | 35
Completed | 36 | 31
Not Completed | 0 | 4
Not completed — Adverse Event | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HQ® Matrix Medical Wound Dressing | Sidaiyi® Wound Dressing | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.39 (14.29) | 37.80 (14.73) | 37.59 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 26
  Male | 26 | 19 | 45

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Growth of Granulation Tissue
Description: Physician assessment of tissue with healthy granulation tissue defined as is granular and uneven in texture, does not bleed easily and is pink in color. Unhealthy granulation tissue is typically dark which can be indicative of poor perfusion, ischemia and/or infection.
Time Frame: Days 0, 3±1, 7±1, 10±2, 14±3, and 21±3 post-operation
Measure: Number; unit: participants
Arm/Group | HQ® Matrix Medical Wound Dressing | Sidaiyi® Wound Dressing
Number analyzed (Participants) | 36 | 35
participants
  Participants with healthy granulation tissue | 36 | 34
  Participants with unhealthy granulation tissue | 0 | 1
Statistical Analysis 1: Comparison: HQ® Matrix Medical Wound Dressing vs Sidaiyi® Wound Dressing; Two-sided Fisher's exact test was performed to assess statistically significant differences of the data of the Number of Participants with Growth of Granulation Tissue between the group treated with the HQ® Matrix Medical Wound Dressing and that treated with the Sidaiyi® wound dressing. This Statistical Analysis applies to the "Participants with healthy granulation tissue" and the "Participants with unhealthy granulation tissue" category; Test type: Superiority or Other; p = 0.49, Fisher Exact — Values of p < 0.05 were considered to be significantly different

2. Secondary Outcome: Number of Participants With Inflammatory Reaction
Description: Physician assessment determined presence of inflammatory reaction which is characterized by pain, heat, redness and swelling.
Time Frame: Days 0, 3±1, 7±1, 10±2, 14±3, and 21±3 post-operation
Measure: Number; unit: participants
Arm/Group | HQ® Matrix Medical Wound Dressing | Sidaiyi® Wound Dressing
Number analyzed (Participants) | 36 | 35
participants
  Participants with Inflammatory Reaction | 1 | 3
  Participants without Inflammatory Reaction | 35 | 32
Statistical Analysis 1: Comparison: HQ® Matrix Medical Wound Dressing vs Sidaiyi® Wound Dressing; Two-sided Fisher's exact test was performed to assess statistically significant differences of the data of the Number of Participants with Inflammatory Reaction between the group treated with the HQ® Matrix Medical Wound Dressing and that treated with the Sidaiyi® wound dressing. This Statistical Analysis applies to the "Participants with Inflammatory Reaction" and the "Participants without Inflammatory Reaction" category; Test type: Superiority or Other; p = 0.36, Fisher Exact — Values of p < 0.05 were considered to be significantly different

3. Secondary Outcome: Pain Perceived by Patient
Description: The amount of pain that a patient perceived was assessed using a Visual Analogue Scale (VAS 0-10), which ranges across a continuum from 0 (no pain) to 10 (worst pain).
Time Frame: Days 0, 3±1, 7±1, 10±2, 14±3, and 21±3 post-operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HQ® Matrix Medical Wound Dressing | Sidaiyi® Wound Dressing
Number analyzed (Participants) | 36 | 35
units on a scale | 0.75 (0.91) | 1.14 (1.14)
Statistical Analysis 1: Comparison: HQ® Matrix Medical Wound Dressing vs Sidaiyi® Wound Dressing; Two-sided t-test was performed to assess statistically significant differences of the data of the VAS score between the group treated with the HQ® Matrix Medical Wound Dressing and that treated with the Sidaiyi® wound dressing; Test type: Superiority or Other; p = 0.11, t-test, 2 sided — Values of p < 0.05 were considered to be significantly different

4. Secondary Outcome: Number of Participants With Exudation
Description: Physician assessment determined presence of exudation by observing whether the gauze over the primary wound dressings was soaked by exudation:
  1. Less than two gauze was soaked by exudation within 24h---No exudation (-);
  2. Two to four gauze was soaked by exudation within 24h---Little exudation (+);
  3. More than four gauze was soaked by exudation within 24h---Much exudation (++);
Time Frame: Days 0, 3±1, 7±1, 10±2, 14±3, and 21±3 post-operation
Measure: Number; unit: participants
Arm/Group | HQ® Matrix Medical Wound Dressing | Sidaiyi® Wound Dressing
Number analyzed (Participants) | 36 | 35
participants
  No exudation (-) | 36 | 32
  Little exudation (+) | 0 | 3
  Much exudation (++) | 0 | 0
Statistical Analysis 1: Comparison: HQ® Matrix Medical Wound Dressing vs Sidaiyi® Wound Dressing; Two-sided Fisher's exact test was performed to assess statistically significant differences of the data of the Number of Participants with Exudation between the group treated with the HQ® Matrix Medical Wound Dressing and that treated with the Sidaiyi® wound dressing. This Statistical Analysis applies to "No exudation" and "Little exudation" category; Test type: Superiority or Other; p = 0.11, Fisher Exact — Values of p < 0.05 were considered to be significantly different

5. Primary Outcome: Time to Wound Healing
Description: Healing time was recorded when complete re-epithelialization had occurred. If the wound healed in advance, visit until the wound was completely healed. If the wounds were unable to heal for more than 21±3 days, unanticipated follow-ups were added until the wound was completely healed.
Time Frame: Days 0, 3±1, 7±1, 10±2, 14±3, and 21±3 post-operation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | HQ® Matrix Medical Wound Dressing | Sidaiyi® Wound Dressing
Number analyzed (Participants) | 36 | 31
Days | 9.86 (1.79) | 11.35 (3.03)
Statistical Analysis 1: Comparison: HQ® Matrix Medical Wound Dressing vs Sidaiyi® Wound Dressing; Two-sided t-test was performed to assess statistically significant differences of the data of the Time to Wound Healing between the group treated with the HQ® Matrix Medical Wound Dressing and that treated with the Sidaiyi® wound dressing; Test type: Superiority or Other; p = 0.02, t-test, 2 sided — Values of p < 0.05 were considered to be significantly different

ADVERSE EVENTS:
Arm/Group | HQ® Matrix Medical Wound Dressing | Sidaiyi® Wound Dressing
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 0/36 | 4/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HQ® Matrix Medical Wound Dressing (N=36) | Sidaiyi® Wound Dressing (N=35)
Empyema (Skin and subcutaneous tissue disorders) | 0 | 3
Excessive fluid leakage with odors (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days